CLINICAL TRIAL: NCT04410419
Title: In Individuals With Diabetes Undergoing Elective Colorectal Surgery, Is Carbohydrate Loading Preoperatively Safe? A Pilot Randomized Controlled Trial
Brief Title: Carbohydrate Loading and Diabetes in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Carbs Drink in Colorectal
Record Dates: First submitted 2020-05-22; First posted 2020-06-01 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Surgery; Surgery--Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Standard care for patients with diabetes pre-operatively .
- Carbohydrate drink (Experimental): Carbohydrate drink containing 40g of carbohydrate to be consumed three hours prior to surgery
  Interventions: Dietary Supplement: Pre-operative carbohydrate drink

INTERVENTIONS:
Dietary Supplement: Pre-operative carbohydrate drink — Carbohydrate drink containing 40g of carbohydrate to be consumed three hours prior to surgery
  Arms: Carbohydrate drink

SUMMARY:
The goal of this study is to evaluate the feasibility of conducting a large study that would assess the safety of carbohydrate drinks (i.e. juice) prior to elective colorectal surgery in patients with type 2 diabetes.

Traditionally, prior to surgeries involving a general anesthetic, patients have been told not to eat or drink anything after midnight due to the risk of aspiration. More recent research have shown that it is safe to have clear fluids up to 2 hours before an operation and this is reflected in the current anesthesia clinical guidelines. Moreover, it has been shown that subjecting patients to a state of starvation causes stress on the body that may lead to complications such as poor wound healing, infections, and delayed return to bowel function. A sugar drink before surgery has been shown to be beneficial and can lead to decreased complication rates and decreased length of stay after surgery.

However, it is currently not known if it is safe for patients with type 2 diabetes to have a sugar drink before their surgery since they have trouble processing sugars and a subset of patients with diabetes are at increased risk of aspiration due to delayed stomach emptying.

This feasibility study is designed to answer the question of whether a large scale trial can be conducted examining the benefits of a pre-operative sugar drink in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* All adult (>=18 years of age) patients with an established diagnosis of type 2 diabetes mellitus undergoing elective colorectal surgery at the University of Alberta Hospital, the Grey Nuns Hospital, the Royal Alexandra Hospital or the Misericordia Hospital will be eligible. Only patients treated with diet or oral hypoglycemic agents will be included.

Exclusion Criteria:

* Subjects <18 years of age, and those on insulin therapy preoperatively will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mean difference of preoperative glucose between the two groups | Pre-operative
  Examined in a non-inferiority fashion with NI margin set as 2mmol/L

SECONDARY OUTCOMES:
Composite outcome of diabetes-related complications | Within 30 days of surgery or to discharge
  hypoglycemia, DKA, cancellation of surgery, ketosis or perioperative aspiration
length of stay | Within 30 days of surgery or to discharge
  How long the patient stays in hospital after surgery in days
Surgical site infection | Within 30 days of surgery or to discharge
  Whether a wound infection is noted in hospital
Postoperative complications using the Clavien Dindo scale | Within 30 days of surgery or to discharge
  A composite measure of post-operative complications stratified based on the Clavien Dindo scale from 1-5 with increasing severity from 1 to 5.
Post-operative serum blood glucose concentration | Within 30 days of surgery or to discharge
  Serum blood glucose compiled on a daily basis
Rate of peri-operative insulin use | Within 30 days of surgery or to discharge
  Whether insulin or an insulin infusion in the peri-operative period is used

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No